CLINICAL TRIAL: NCT03794258
Title: A Phase 2a, Open-label, Randomized Study of the Safety and Preliminary Efficacy of Triple or Quadruple Combination DAAs With Ultra-short Duration Therapy in Subjects With HCV Genotype 1b Infection (YANGTZE Study)
Brief Title: Triple or Quadruple Combination DAAs Treatment for Subjects With HCV GT 1b Infection
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Can not recruit the patients due to the pandemic of COVID-19
Sponsor: Humanity & Health Medical Group Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H&H_YANGTZE_1
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: HCV Infection
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SOF+DCV+CDI-31244 (Experimental): Subjects will receive two weeks of sofosbuvir, daclatasvir, and CDI-31244 if they achieve HCV RNA < 500 IU/mL on Day 2 and HCV RNA < LLOQ (< 25 IU/mL) on Week 1.
  Interventions: Drug: SOF+DCV+CDI-31244
- SOF+DCV+CDI-31244+ASV (Experimental): Subjects will receive two weeks of sofosbuvir, daclatasvir, CDI-31244 and asunaprevir if they achieve HCV RNA < 500 IU/mL on Day 2 and HCV RNA < LLOQ (< 25 IU/mL) on Week 1.
  Interventions: Drug: SOF+DCV+CDI-31244+ASV

INTERVENTIONS:
Drug: SOF+DCV+CDI-31244 — Sofosbuvir (SOF) 400 mg administered orally once daily; Daclatasvir (DCV) 60 mg administered orally once daily; CDI-31244 400 mg administered orally once daily.
  Arms: SOF+DCV+CDI-31244
Drug: SOF+DCV+CDI-31244+ASV — Sofosbuvir (SOF) 400 mg administered orally once daily; Daclatasvir (DCV) 60 mg administered orally once daily; CDI-31244 400 mg orally once daily; Asunaprevir (ASV) 200mg administered orally twice daily.
  Arms: SOF+DCV+CDI-31244+ASV

SUMMARY:
This is a phase 2a, open-label, randomized study. The study is designed to test the hypothesis that the nucleoside inhibitor sofosbuvir combined with NS5A inhibitor daclatasvir and NS5B non-nucleoside inhibitor CDI-31244 with/without the protease inhibitor asunaprevir will result in high SVR rate with a shortened treatment duration (2 weeks) in non-cirrhotic HCV genotype 1b-infected subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Male or female, age 18-70 years.
3. HCV genotype 1b infection as determined by the Laboratory. Any non-definitive results will exclude the subject from study participation.
4. HCV RNA level ≥ 10,000 IU/mL and < 10,000,000 IU/mL.
5. No evidence of cirrhosis. Cirrhosis defined as any 1 of the following, within 6 months of study entry:

   1. Liver biopsy showing cirrhosis;
   2. Fibroscan showing cirrhosis or results >12.5 kPa;
   3. FibroTest® score >0.75 and an aspartate aminotransferase (AST): platelet ratio index (APRI) >2 during screening.
6. Subjects must have the following laboratory parameters at screening:

   1. ALT ≤ 10 x the upper limit of normal (ULN);
   2. AST ≤ 10 x ULN;
   3. Direct bilirubin ≤1.5 x ULN;
   4. Platelets ≥ 50,000;
   5. HbA1c ≤ 8.5%;
   6. Creatinine clearance (CLcr) ≥ 60 mL /min, as calculated by the Cockcroft-Gault equation;
   7. Hemoglobin ≥ 11 g/dL for female subjects; ≥ 12 g/dL for male subjects;
   8. Albumin ≥ 3g/dL;
   9. INR ≤ 1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR.
7. Subject has not been treated with any investigational drug or device within 30 days of the Screening visit.
8. A female subject is eligible to enter the study if it is confirmed that she is:

   1. Not pregnant or nursing;
   2. Of non-childbearing potential (i.e., women who have had a hysterectomy, have both ovaries removed or medically documented ovarian failure, or are postmenopausal - women > 50 years of age with cessation (for ≥12 months) of previously occurring menses), or
   3. Of childbearing potential (i.e., women who have not had a hysterectomy, both ovaries removed, or no medically documented ovarian failure) based on the following conditions.

   Women ≤ 50 years of age with amenorrhea will be considered to be of childbearing potential. These women must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on the Baseline/Day 0 visit prior to randomization. They must also agree to one of the following from 3 weeks prior to Baseline/Day 0 until 4 months after last dose of the triple/quadruple therapies:

   - Complete abstinence from intercourse. Periodic abstinence from intercourse (e.g., calendar, ovulation, symptothermal, post-ovulation methods) is not permitted.

   Or
   * Consistent and correct use of 1 of the following methods of birth control listed below in addition to a male partner who correctly uses a condom from 3 weeks prior to Baseline/Day 0 until 4 months after last dose of the triple/quadruple therapies. Women of childbearing potential must not rely only on hormone-containing contraceptives as a form of birth control during the study. Female subjects using a hormone-containing contraceptive prior to Screening may continue their contraceptive regimen in addition to the study specified methods of birth control.
   * intrauterine device (IUD) with a failure rate of <1% per year
   * female barrier method: cervical cap or diaphragm with spermicidal agent
   * tubal sterilization
   * vasectomy in male partner
9. All male study participants must agree to consistently and correctly use a condom, while their female partner agrees to use either 1 of the non-hormonal methods of birth control listed above or a hormone-containing contraceptive listed below, from the date of Screening until 4 months after their last dose of the triple/quadruple therapies:

   * implants of levonorgestrel
   * injectable progesterone
   * oral contraceptives (either combined or progesterone only)
   * contraceptive vaginal ring
   * transdermal contraceptive patch
10. Male subjects must agree to refrain from sperm donation from the date of screening until at least 4 months after the last dose of the triple therapies.
11. Subject must be of generally good health, with the exception of chronic HCV infection, as determined by the Investigator.
12. Subject must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments.
13. Screening ECG without clinically significant abnormalities.

Exclusion Criteria:

1. Child-Pugh scoring of B and C.
2. Creatinine Clearance < 30ml/min.
3. Mixed HCV genotypes.
4. Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV).
5. Hepatocellular carcinoma or other malignancy (with exception of certain resolved skin cancers).
6. Current or prior history of any of the following:

   1. Clinically-significant illness (other than HCV) or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol; subjects currently under evaluation for a potentially clinically-significant illness (other than HCV) are also excluded.
   2. Gastrointestinal disorder or post operative condition that could interfere with the absorption of the study drug.
   3. Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy.
   4. Clinical hepatic decompensation (i.e., ascites, encephalopathy or variceal hemorrhage).
   5. Solid organ transplantation.
   6. Significant pulmonary disease, significant cardiac disease or porphyria.
   7. Psychiatric hospitalization, suicide attempt, and/or a period of disability as a result of their psychiatric illness within the last 5 years. Subjects with psychiatric illness that is well-controlled on a stable treatment regimen for at least 12 months prior to randomization or has not required medication in the last 12 months may be included.
   8. Malignancy diagnosed or treated within 5 years (recent localized treatment of squamous or non-invasive basal cell skin cancers is permitted; cervical carcinoma in situ is allowed if appropriately treated prior to screening); subjects under evaluation for malignancy are not eligible.
   9. Significant drug allergy (such as anaphylaxis or hepatotoxicity).
   10. History or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the subject's participation for the full duration of the study, such that it is not in the best interest of the subject to participate
7. Pregnant or nursing female or male with pregnant female partner.
8. Chronic liver disease of a non-HCV etiology (e.g., hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, cholangitis).
9. Donation or loss of more than 400 mL blood within 2 months prior to Baseline/Day 1.
10. Clinically-relevant drug abuse within 12 months of screening. A positive drug screen will exclude subjects unless it can be explained by a prescribed medication; the diagnosis and prescription must be approved by the investigator.
11. Active or recent history (≤ 1 year) of drug or alcohol abuse.
12. Use of any following drugs that might interact with the study drugs.

    1. Treatment with amiodarone within 180 days before study entry;
    2. Treatment with digoxin within 30 days before study entry;
    3. Treatment with rifabutin, rifampin, rifapentine, phenytoin, phenobarbital, St. John's wort, carbamazepine, oxcarbazepine, rosuvastatin, or atorvastatin within 10 days before study entry. However, switching to another statin is acceptable.
13. Screening or baseline electrocardiogram (ECG) with clinically significant findings.
14. QTcF (QT interval corrected using Fridericia's formula) > 450 msec at screening.
15. Chronic use of systemically administered immunosuppressive agents (e.g., prednisone equivalent > 10 mg/day).
16. Known hypersensitivity to sofosbuvir, daclatasvir, CDI-31244 and asunaprevir or formulation recipients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with sustained virologic response 12 weeks after discontinuation of therapy (SVR12) | Post treatment Week 12
  SVR12 is defined as HCV RNA < lower limit of quantification (LLOQ) 12 weeks after last dose of study drug.

SECONDARY OUTCOMES:
Frequency and severity of adverse events | Baseline up to Week 24
Proportion of participants with unquantifiable HCV viral load at specified time points during and after treatment | Baseline up to Week 24
HCV RNA levels and change during and after treatment | Baseline up to Week 24
Proportion of participants with on-treatment virologic breakthrough and relapse | Baseline up to Week 24
  Viral breakthrough is defined as having achieved undetectable HCV RNA levels (HCV RNA < LLOQ) during treatment, but did not achieve a sustained virologic response (SVR). Viral relapse is defined as having achieved undetectable HCV RNA levels (HCV RNA < LLOQ) within 4 weeks of end of treatment, but did not achieve an SVR.

CONTACTS AND LOCATIONS:
Overall Officials: Georg Lau, MD, Principal Investigator — Humanity & Health Research Centre
Locations (1):
- Humanity & Health Research Centre, Hong Kong, Hong Kong SAR, Hong Kong